CLINICAL TRIAL: NCT07270614
Title: Effects of an 8-Week Injury Prevention Program on Lower Limb Performance in Female Athletes: Quasi-Experimental Evidence
Brief Title: Eight-week Sports Injury Prevention Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Sponsor-Investigator, Princess Nourah Bint Abdulrahman University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PNU-7
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Health Adult Subjects
Keywords: Injury prevention program

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): Participants will attend supervised injury-prevention sessions for eight weeks. Each session includes:
  Warm-up drills (jogging, shuttle runs, backward running)
  Stretching for major lower-body muscles
  Strength training such as lunges and hamstring exercises
  Plyometric drills (jumping and bounding)
  Balance exercises on one leg
  Agility drills such as directional running
  Cool-down stretching and core exercises
  This type of program is commonly used to reduce lower-limb injuries by improving strength, stability, coordination, and movement control.
  Interventions: Behavioral: 8-Week Sports Injury Prevention Program

INTERVENTIONS:
Behavioral: 8-Week Sports Injury Prevention Program — A structured 8-week injury prevention exercise program designed to improve lower-extremity strength, balance, agility, and movement control in female college athletes. Each supervised session includes:
  Warm-up: jogging, shuttle runs, backward running
  Stretching: calf, quadriceps, and hamstring stretches
  Strengthening: walking lunges, Russian hamstring exercise, single-leg toe raises
  Plyometrics: lateral, forward, and backward jumps; zigzag shuffle; bounding drills
  Balance training: single-leg stance with chest pass, forward bend, and figure-of-eight reach
  Agility drills: multidirectional shuttle runs, diagonal runs, bounding runs
  Cool-down: bridging, abdominal crunches, knee-to-chest stretches, and seated butterfly stretch
  Sessions follow a standardized protocol with prescribed repetitions, sets, or time durations for each component. The goal of the intervention is to enhance athletic performance and reduce the risk of lower-extremity sports injuries.

SUMMARY:
This study aims to find out whether an 8-week sports injury prevention program can improve lower-body performance-such as power, agility, and balance-among female college athletes in Saudi Arabia.

Sports participation has increased among women in Saudi Arabia, but many injury-prevention programs were originally designed for male athletes and may not meet the specific needs of females. This study will help determine whether a tailored program can reduce injury risks and improve athletic performance.

Female athletes aged 18-35 years who have been training and competing for at least one year can participate. Athletes with recent injuries, pregnancy, or chronic medical conditions that could affect performance will not be included.

Participants will complete tests before and after the program, including jumping, balance, and agility assessments. The prevention program includes warm-up exercises, stretching, strengthening, jumping drills, balance work, and agility training.

By comparing results before and after the program, the study will show whether this type of training can help female athletes stay safer and perform better.

DETAILED DESCRIPTION:
This study will evaluate whether an 8-week sports injury prevention program can improve injury-related knowledge and lower-body performance in female college athletes. Sports participation among women in Saudi Arabia has increased in recent years, but female athletes often use injury-prevention programs originally designed for men. Because women have different physical and biomechanical characteristics, they may face a higher risk of sports injuries. This study aims to address this gap by testing a program tailored to their needs.

Participants will attend supervised injury-prevention sessions for eight weeks. Each session includes:

Warm-up drills (jogging, shuttle runs, backward running)

Stretching for major lower-body muscles

Strength training such as lunges and hamstring exercises

Plyometric drills (jumping and bounding)

Balance exercises on one leg

Agility drills such as directional running

Cool-down stretching and core exercises

This type of program is commonly used to reduce lower-limb injuries by improving strength, stability, coordination, and movement control.

How participation will be assessed

Before starting the program and again after the eight weeks, participants will complete several tests that measure:

Jumping power

Agility during multi-directional movement

Balance while reaching in different directions

These tests are widely used in sports medicine and have high reliability. They help identify injury risk and measure improvements in physical performance.

Why this study is important

The results will show whether a structured injury-prevention program can help female athletes:

Improve movement quality

Enhance lower-body strength, balance, and agility

Increase awareness of sports-injury risks

Potentially reduce the likelihood of future injuries

This research may support the development of safer and more effective training strategies for female athletes in Saudi Arabia as sports opportunities continue to expand.

ELIGIBILITY:
Inclusion Criteria:

* Female athletes aged 18-35 years
* Actively participating in organized sports in Saudi Arabia
* Minimum of one year of continuous experience in their sport
* Currently engaged in regular training and/or competition
* Able to perform physical activity safely as confirmed by self-report
* Willing to provide informed consent and complete all study assessments

Exclusion Criteria:

* Any recent injury within the past six months that limits performance
* Pregnancy at the time of enrollment
* Diagnosis of a chronic medical condition that may affect performance (e.g., uncontrolled diabetes, uncontrolled hypertension)
* Any condition that could interfere with safe participation in physical testing or training
* Refusal or inability to provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-16 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Lower-Extremity Functional Performance | From enrollment to the end of treatment at 8 weeks
  Description: Assessed using the Lower Extremity Functional Test (LEFT), which evaluates multidirectional agility through eight standardized tasks (forward run, backward run, side shuffle, carioca, figure-8 run, 45° cuts, 90° cuts, and countermovement jump).
  Time Frame: Baseline and 8 weeks (post-intervention). Outcome Metric: Total completion time (seconds). Lower times indicate better performance.
Change in Lower-Body Explosive Power | From enrollment to the end of treatment at 8 weeks
  Description: Measured using the Countermovement Jump (CMJ) and Standing Long Jump (SLJ) tests, both widely validated for assessing lower-limb power.
  Time Frame: Baseline and 8 weeks. Outcome Metric: CMJ height (cm) and SLJ distance (cm).
Change in Dynamic Balance | From enrollment to the end of treatment at 8 weeks
  Description: Evaluated using the Star Excursion Balance Test (SEBT) in the anterior, posteromedial, and posterolateral directions.
  Outcome Metric: Max reach distance (cm), normalized to leg length.

CONTACTS AND LOCATIONS:
Locations (1):
- PNU- Students gym, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided